CLINICAL TRIAL: NCT01688375
Title: The Effect of Ursodeoxycholic Acid in Liver Functional Restoration of Patients With Obstructive Jaundice After Endoscopic or Surgical Treatment
Brief Title: The Effect of Ursodeoxycholic Acid in Liver Functional Restoration of Patients With Obstructive Jaundice
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Clinical Centre of Kosova (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Principal Investigator, Enver Fekaj, General surgeon, PhD student, University Clinical Centre of Kosova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E25071969F; EN1969FE (Other: University clinical centre of Kosovo)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Obstructive Jaundice
Keywords: obstructive jaundice; ursodeoxycholic acid
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ursodeoxycholic acid (Experimental): Ursodeoxycholic acid administration UDCA administration will begin twenty-four hours after endoscopic or surgical procedure and will last fourteen days. UDCA dose will be administered at 750 mg/day, divided into three doses.
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — UDCA administration will begin twenty-four hours after endoscopic or surgical procedure and will last fourteen days. UDCA dose will be administered at 750 mg/day, divided into three doses.
  Other Names: Ursofalk, UDCA

SUMMARY:
ABSTRACT:

In patients with obstructive jaundice, multi-organ dysfunction may develop. The aim of this study is to evaluate the effect of ursodeoxycholic acid on liver functional restoration on patients with obstructive jaundice after surgical or endoscopic treatment.

Patients with obstructive jaundice will be divided into two groups: (A) test group in which will be administered ursodeoxycholic acid twenty-four hours after endoscopic or surgical procedure and will last fourteen days, and (B) control group.

Serum-testing will include determination of bilirubin, alanine transaminase, aspartate transaminase, gama-glutamyl transpeptidase, alkaline phosphatase, albumin, and cholesterol levels. These parameters will be determined one day prior endoscopic or surgical procedure, and on the third, fifth, seventh, tenth, twelfth and fourteenth days after endoscopic or surgical intervention.

Our hypothesis is that patients with obstructive jaundice under treatment with ursodeoxycholic acid will have better outcome than patients in control group.

DETAILED DESCRIPTION:
Study objectives:

This trial will be a prospective, an open, randomized and controlled study. The objective will be to evaluate the effect of ursodeoxycholic acid (UDCA) in the functional restoration of the liver in patients with obstructive jaundice in the early post-endoscopic or post-surgical phase.

Study design:

After diagnosis, patients with obstructive jaundice will be divided into two groups: (A) the test group in which will be administered UDCA in the early phase after endoscopic or surgical treatment, and (B) control group, in which no treatment will be applied with UDCA.

Diagnostic methods will be biochemical findings, ultrasound examination, endoscopic retrograde cholangio pancreatography (ERCP), CT-scan and magnetic resonance cholangio pancreatography (MRCP).

Serum-testing in patients with obstructive jaundice will include determination of bilirubin (total and direct fractions), alanine transaminase (ALT), aspartate transaminase (AST), gama-glutamyl transpeptidase (GGT), alkaline phosphatase, albumin, and cholesterol levels. These parameters will be determined one day prior endoscopic or surgical intervention, and on the third, fifth, seventh, tenth, twelfth and fourteenth days after endoscopic or surgical intervention.

Endoscope and surgical procedures that will end with the external derivation of bile will be named as the external bile drainage, and indeed, while endoscope and surgical procedures that will make the internal derivation of bile shall be named as the internal bile drainage.

UDCA administration:

UDCA administration will begin twenty-four hours after endoscopic or surgical procedure and will last fourteen days. UDCA dose will be administered at 750 mg/day, divided into three doses.

Power of the study:

A clinically relevant improvement of liver functional tests is defined as an improvement of 80% of liver functional tests in test group, and an improvement only 40% in control group. In our study, to have an 80% chance of detecting a 50% difference between two groups on improvement of liver functional tests at an alpha level of 0.05, the power calculation indicates that each of the two groups should have at least 27 patients.

Data sources and search strategy:

An electronic search was performed on PubMed (from 1 January 1985 to 1 February 2012). A combination of keywords and MeSH terms where: 'ursodeoxycholic acid' AND 'obstructive jaundice', 'obstructive jaundice' AND 'liver function tests', 'obstructive jaundice' AND 'acute renal failure'. I have used , also, limits: Type of article ( selection was- clinical trial, meta-analyses), Species( selection was- human, animals), Text options ( selection was- links to free full text, abstract), Languages( English), Sex ( male, female), Age ( all adult 19+ years), Field ( all fields).

Randomization:

Patients have to sign an informed consent for the involving in the trial a day before endoscopic or surgical procedure. Randomisation will be performed at the time of transfer to the endoscope or operating room.

Ethics:

This study will be realized in the Surgery Clinic (Department of Abdominal Surgery) at University Clinical Centre of Kosovo in Pristina. It will be conducted in accordance with the principles of the Declaration of Helsinki. This study will begin after approval of the study protocol by Medical Ethics Committee of the University Clinical Centre of Kosovo( Faculty of Medicine).

Data collection and statistical analyses:

Data including serum-test results will be collected in a computer secured study platform. These data will be collected continuously, for each patient, starting one day before endoscopic or surgical procedure until the last data fourteen days after intervention.

X2-analysis or Fisher exact test will perform to test the differences in proportions of qualitative variables between groups. Mann Whitney U test and Kruskal Wallis test will use for testing the difference between quantitative variables when distribution is not normal and Student t-test or ANOVA test when distribution is normal. The level P<0.05 will consider as the cut-off value for significance.

ELIGIBILITY:
Inclusion criteria:

* Patients with obstructive jaundice
* Serum bilirubin level higher than 50 micromole/l
* 19+ years of age
* written informed consent

Exclusion criteria:

* Cholangitis
* Acute pancreatitis
* pregnant women
* women during the breastfeeding
* suspected or proven primary liver diseases
* My family members
* Patients who are unable to understand our study purpose

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Liver functional restoration | Within 14 days after treatment with ursodeoxycholic acid
  Serum-testing in patients with obstructive jaundice will include determination of bilirubin (total and direct fractions), alanine transaminase (ALT), aspartate transaminase (AST), gama-glutamyl transpeptidase (GGT), alkaline phosphatase, albumin, and cholesterol levels.

SECONDARY OUTCOMES:
To assess that in which functional parameters of the liver, treatment with UDCA will have greater impact | within 14 days after treatment with ursodeoxycholic acid
  determination of bilirubin (total and direct fractions), alanine transaminase (ALT), aspartate transaminase (AST), gama-glutamyl transpeptidase (GGT), alkaline phosphatase, albumin, and cholesterol levels. These parameters will be determined one day prior endoscopic or surgical intervention, and on the third, fifth, seventh, tenth, twelfth and fourteenth days after endoscopic or surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Enver H Fekaj, PhD student, Principal Investigator — University clinical centre of Kosovo, Department of surgery
Locations (2):
- Serbia (2):
  - University clinical centre of Kosovo, Department of general surgery, Pristina, Kosovo
  - University clinical centre of Kosovo, Pristina, Kosovo

REFERENCES:
- [Background] 1. Roche SP, Kobos R. Jaundice in the adult patient. Am Fam Physician. 2004; 69(2):299-304. 2. Rerknimitr R, Kullavanijaya P. Operable malignant jaundice: To stent or not to stent before the operation? World J Gastrointest Endosc. 2010; 2(1):10-4. 3.Yi-Jun Y, Jing-Sen SH, Shu-Min X, De-Ting ZH, Bing-Sheng C. Effects of different drainage procedures on levels of serum endotoxin and tumor necrosis factor in patients with malignant obstructive jaundice. HBPD Int. 2003;2:426-30. 4.Scott-Conner CE, Grogan JB. The pathophysiology of biliary obstruction and its effect on phagocytic and immune function. J Surg Res. 1994;57(2):316-36. 5.Assimakopoulos SF, Scopa ChD, Vaginos CE. Pathophysiology of increased intestinal permeability in obstructive jaundice. World J Gastroenterol. 2007;13(48):6458-64.
- [Derived] Fekaj E, Gjata A, Maxhuni M. The effect of ursodeoxycholic acid in liver functional restoration of patients with obstructive jaundice after endoscopic treatment: a prospective, randomized, and controlled study. BMC Surg. 2013 Sep 22;13:38. doi: 10.1186/1471-2482-13-38. PMID 24053627